CLINICAL TRIAL: NCT00837694
Title: Differential Effects of Daily Snack Food Intake on Reinforcing Value of Food in Obese and Non-obese Women.
Brief Title: Snack Food Reinforcement in Obese and Non-obese Women
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jennifer Temple, Assistant Professor, State University of New York at Buffalo
Other Study IDs: Temple1
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: BMI; obesity; sensitization; food reinforcement; snack food; Portion size of daily snacks; Weight status
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Non-obese/0 kcal
- 2: Non-obese/100 kcal
- 3: Non-obese/300 kcal
- 4: Obese/0 kcal
- 5: Obese/100 kcal
- 6: Obese/300 kcal

SUMMARY:
Food reinforcement, motivation to obtain food, is associated with energy intake and obesity. Finding ways to decrease the reinforcing value of unhealthy foods may help with adherence to diets and weight loss. Our previous study in non-obese adults showed that daily consumption of the same snack food (food typically consumed outside of meals) for 14 days significantly decreased its reinforcing value. The purpose of this study was to replicate and extend these findings to obese individuals as well as to examine effects of different portion sizes of snack foods on food reinforcement. Thirty-one obese (body mass index > 30 kg/m2) and 27 non-obese (BMI < 30 kg/m2) women had food reinforcement and liking tested at baseline and after two weeks of daily consumption of either 0 kcal, 100 kcals, or 300 kcals daily of the same snack food.

ELIGIBILITY:
Inclusion Criteria:

* women
* non-smoker
* not on a diet
* no restrained eating
* had to like potential snack foods
* willing to visit the laboratory 3 times
* willing to eat snacks provided
* no medications or medical conditions that affect appetite
* no food allergies

Exclusion Criteria:

* see above

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women ages 18 - 50 years who were obese (body mass index >/= 30) or non-obese (BMI < 30)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Temple, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Temple JL, Bulkley AM, Badawy RL, Krause N, McCann S, Epstein LH. Differential effects of daily snack food intake on the reinforcing value of food in obese and nonobese women. Am J Clin Nutr. 2009 Aug;90(2):304-13. doi: 10.3945/ajcn.2008.27283. Epub 2009 May 20. PMID 19458018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from flyers poster around campus. Interested participants called the lab and were screened by telephone.
Pre-assignment Details: Exclusionary criteria included smoking, current dieting, medications that could affect appetite, medical conditions that limited physical activity, allergies to or self-reported dislike of study foods.
Groups:
- Non-Obese/0 kcal: Non-obese participants that received no snack food to consume for two weeks.
- Non-Obese/100 kcal: Non-obese participants that received a 100 kcal portion of food to consume daily for two weeks.
- Non-obese/300 kcal: Non-obese participants that received a 300 kcal portion of food to consume daily for two weeks.
- Obese/0 kcal: Obese participants that received no food to consume for two weeks.
- Obese/100 kcal: Obese participants that received a 100 kcal portion of food to consume daily for two weeks.
- Obese/300 kcal: Obese individuals who received a 300 kcal portion of food to consume for 2 weeks.
Period: Overall Study
Arm/Group | Non-Obese/0 kcal | Non-Obese/100 kcal | Non-obese/300 kcal | Obese/0 kcal | Obese/100 kcal | Obese/300 kcal
Started | 10 | 11 | 10 | 11 | 12 | 11
Completed | 8 | 11 | 8 | 10 | 11 | 10
Not Completed | 2 | 0 | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Obese/0 kcal | Non-Obese/100 kcal | Non-obese/300 kcal | Obese/0 kcal | Obese/100 kcal | Obese/300 kcal | Total
Number analyzed (Participants) | 10 | 11 | 10 | 11 | 12 | 11 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 10 | 11 | 12 | 11 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.57 (7.37) | 26.57 (9.49) | 29.13 (7.37) | 31.4 (2.69) | 37.82 (2.85) | 38.79 (3.72) | 32.13 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 11 | 12 | 11 | 65
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Race (minority/non-minority)
  participants
    Minority | 1 | 1 | 2 | 6 | 4 | 3 | 17.0
    Non-Minority | 9 | 10 | 8 | 5 | 8 | 8 | 48.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Responses Made by Clicking a Mouse Button for Food
Description: Participants were asked to click a button on a computer mouse and after a certaion number of responses, participants would receive a point. After 5 points, the participants received a portion of snack food.
Time Frame: During 2nd and 3rd visits
Measure: Mean (Standard Error); unit: Number of button presses
Arm/Group | Non-Obese/0 kcal | Non-Obese/100 kcal | Non-obese/300 kcal | Obese/0 kcal | Obese/100 kcal | Obese/300 kcal
Number analyzed (Participants) | 8 | 11 | 8 | 10 | 11 | 10
Number of button presses
  Number of responses at baseline | 397.63 (307.6) | 288.36 (68.44) | 429.5 (307.7) | 213.2 (72.51) | 448.36 (217.49) | 502.00 (257.05)
  Number of responses visit 3 | 170.38 (77.48) | 227.27 (50.80) | 115.25 (46.82) | 147.2 (27.23) | 468.18 (298.40) | 1063.6 (670.32)

2. Primary Outcome: Energy Intake
Description: energy contained in eaten foods and beverages
Time Frame: visits 1, 2, and 3 plus on the phone throughout the study.
Reporting Status: Not Posted

3. Secondary Outcome: Body Weight
Description: body weight
Time Frame: visit 1 and visit 3
Reporting Status: Not Posted

4. Secondary Outcome: Height
Description: height
Time Frame: visits 1 and 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Non-Obese/0 kcal | Non-Obese/100 kcal | Non-obese/300 kcal | Obese/0 kcal | Obese/100 kcal | Obese/300 kcal
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/11 | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
One limitation was that we relied on self-report for energy and snack food intake. It is possible that people were not eating the food that they said they were. Another limitation was that people may have not understood the task.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes